CLINICAL TRIAL: NCT05345509
Title: A Phase 1, Randomized, Open-Label, Exploratory, Sequential, Pharmacokinetic Single Ascending Dose Study of IVL3003 Versus Multiple Doses of Aricept (Donepezil) Tablets in Healthy Subjects
Brief Title: A Clinical Trial to Access Pharmacokinetic Profiles and Safety of IVL3003.
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inventage Lab., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IVL3003-001
Record Dates: First submitted 2022-04-19; First posted 2022-04-26 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Aricept Tablet (Active Comparator): Aricept Tablet, QD, PO
  Interventions: Drug: Aricept Tablet
- IVL3003 (A mg) (Experimental): SC, Single Dose
  Interventions: Drug: IVL3003
- IVL3003 (B mg) (Experimental): SC, Single Dose
  Interventions: Drug: IVL3003
- IVL3003 (C mg) (Experimental): SC, Single Dose
  Interventions: Drug: IVL3003
- IVL3003 (Dmg) (Experimental): Intramuscular
  Interventions: Drug: IVL3003
- IVL3003 (Emg) (Experimental): Intramuscular
  Interventions: Drug: IVL3003

INTERVENTIONS:
Drug: Aricept Tablet — Donepezil Tablet once daily P.O
  Arms: Aricept Tablet
Drug: IVL3003 — Donepezil Long-Acting Injection, once S.C Injection
  Arms: IVL3003 (A mg); IVL3003 (B mg); IVL3003 (C mg)
Drug: IVL3003 — Donepezil Long-Acting Injection, once IM Injection
  Arms: IVL3003 (Dmg); IVL3003 (Emg)

SUMMARY:
A Clinical Trial to Assess Pharmacokinetic Profiles and Safety of IVL3003

DETAILED DESCRIPTION:
A Phase 1, Randomized, Open-Label, Exploratory, Sequential, Pharmacokinetic Single Ascending Dose Study of IVL3003 Versus Multiple Doses of Aricept (Donepezil) Tablets in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female, ≥18 and ≤55 years of age, non-smokers or occasional smokers (defined as smoking less than 10 cigarettes or nicotine equivalent per week, and willing to abstain from smoking during confinement at the study site).
* Body mass index (BMI) ≥18.0 and ≤32.0 kg/m2 and body weight ≥55.0 kg for males and ≥50.0 kg for females.
* Male subjects who are sexually active with a same-sex partner must be willing to use a condom until study exit.
* Male and female subjects who practice abstinence from sexual intercourse as a usual and preferred lifestyle.
* Willing to abstain from use of non-steroidal anti-inflammatory drugs (NSAIDs) including ibuprofen, naproxen, aspirin, meloxicam, etc. from screening until study exit.
* Willing and able to provide written informed consent after the nature of the study has been explained and prior to the commencement of any protocol specific study procedures.

Exclusion Criteria:

* Any clinically significant abnormal finding at physical examination at screening.
* Clinically significant abnormal laboratory test results or positive serology test results for human immunodeficiency virus (HIV), hepatitis B or hepatitis C virus at screening.
* Positive pregnancy test at screening or Day -1 or lactating female subject.
* Positive drug or alcohol screen at screening or Day -1.
* Any history of malignancy or neoplastic disease.
* History of significant allergic reactions (e.g., drug reaction, anaphylactic reaction, hypersensitivity, angioedema) to donepezil, piperidine derivatives, dimenhydrinate or derivatives, benzatropine or derivatives, or other related drugs, or to any excipient present in the formulation for any study drug.
* Presence of hereditary disorders including galactose intolerance, lactase deficiency, and glucose-galactose malabsorption (for Part B only).
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin >1.5x the upper limit of normal (ULN) at screening or Day -1.
* Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2 as calculated by the 2021 Chronic Kidney Disease-Epidemiology (CKD-EPI) equation at screening or Day -1.
* Clinically significant ECG abnormalities (QTc >450 ms or PR interval >220 ms) or vital sign abnormalities (systolic blood pressure <90 or >140 mmHg, diastolic blood pressure <40 or >90 mmHg, or heart rate <50 or >100 bpm) at screening or Day 1.
* History of significant bradycardia or atrioventricular (AV) block.
* History of significant asthma (except for fully resolved childhood asthma) or chronic obstructive pulmonary disease (COPD).
* History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 14 units of alcohol per week (1 unit = 375 mL of beer 3.5%, 100 mL of wine 13.5%, or 30 mL of spirit 40%).
* History of drug abuse within 1 year prior to screening or recreational use of soft drugs (such as marijuana) or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 1 month, or use of codeine within 3 months prior to screening.
* Donation of plasma within 7 days prior to dosing or donation or loss of 500 mL or more of whole blood within 30 days prior to dosing.
* Consumption of high levels of caffeine (equivalent to 3 regular cups of coffee or 2 energy drinks, per day).
* Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-11-13 (Estimated); Study Completion 2025-11-13 (Estimated)

PRIMARY OUTCOMES:
AUClast of IVL3003 | Pre-dose, up to 1month
  Area under the concentration-time curve from time zero to last
AUCinf of IVL3003 | Pre-dose, up to 1month
  Area under the concentration-time curve from time zero to infinity
AUClast of Aricept | Pre-dose, up to 1month
  Area under the concentration-time curve from time zero to last
AUCinf of Aricept | Pre-dose, up to 1month
  Area under the concentration-time curve from time zero to infinity

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No